CLINICAL TRIAL: NCT00670852
Title: Computed Tomographic and Functional Follow-up of Glenoid Anchor Peg Component Fixation Utilizing Autologous Bone Graft in Total Shoulder Arthroplasty
Brief Title: Followup of Glenoid Fix Utilizing Auto Bone Graft in Shoulder Replacement
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0391-07-FB
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Arthritis
Keywords: Glenoid component; radiolucent lines; Glenoid loosening; glenohumeral arthritis; autologous bone graft
MeSH Terms: conditions — Arthritis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total shoulder replacement with anchor peg glenoid and autologous bone grafting: Patients who received a total shoulder replacement with an anchor peg glenoid and autologous bone grafting from the investigator of this study will be recruited for this study.
  Interventions: Procedure: X-rays and CT scan

INTERVENTIONS:
Procedure: X-rays and CT scan — CT Scan x-rays
  Other Names: No names

SUMMARY:
This is a case study to evaluate the adequacy of fixation and functional outcome of the glenoid anchor peg following autologous bone grafting around the prosthesis at the time of implant.

DETAILED DESCRIPTION:
To investigate if the use of autologous bone graft around the anchor-peg glenoid prosthesis correlates with bony apposition on computed tomography scans, decreased radiolucent lines and component loosening, and functional outcomes. We hypothesize that by utilizing autologous bone graft from the resected humeral head, placed around the anchor peg glenoid prosthesis at implantation, there is a low incidence of glenoid loosening. We suggest that the absence of radiolucent lines correlated with excellent shoulder function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a total shoulder replacement with an anchor peg glenoid and autologous bone grafting from the investigator of this study will be recruited for this study.

Exclusion Criteria:

* Patients will be excluded if they are unable to comprehend the consent information.
* Pregnant women will be excluded from this study.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Maximum number will be 70. Patients who received a total shoulder replacement with an anchor peg glenoid and autologous bone grafting from the investigator of this study will be recruited for this study.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2009-06-10 (Actual); Study Completion 2009-06-10 (Actual)

PRIMARY OUTCOMES:
Autologous bone graft, anchor-peg glenoid prosthesis and functional outcomes | case study over approximate 3 months time.
  To determine if the use of autologous bone graft around the anchor-peg glenoid prosthesis correlate with bony apposition on computed tomography scans, decreased radiolucent lines and component loosening, and functional outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Fehringer, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Dept Orthopaedic Surgery, Omaha, Nebraska, United States